CLINICAL TRIAL: NCT05644886
Title: Assessing the Feasibility, Effectiveness and Outcomes of Engaging Family Physicians and Pharmacies to Expand Family Planning Services in Rural Areas of Islamabad
Brief Title: Pilot Study on Engaging Family Physicians in Family Planning in Pakistan
Acronym: FPFP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Population Council (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Ayaz Ahmed Baloch, Program Manager Research, Population Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1014
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Contraceptive Usage; Contraception
Keywords: Family Planning; Pakistan; Family Physicians; Contraceptive; Pharmacies; Male
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: The study uses a two arm parallel facility based randomized controlled trial with on-going intervention of training and technical support for six-month.
Masking Description: Due to the nature of the intervention masking is not feasible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Male Family Physicians allocated to intervention arm will receive following:
  Training and technical support and integrates them with the nearest pharmacies or drug shops for vertical referrals.
  Technical support will include:
  * Supportive supervision
  * Peer-to-peer support
  * Strengthening referrals for long-acting reversible contraceptives (LARC) and permanent methods
  * Provision of information, education, and communication (IEC) material and LCD for display of visual material.
  * Branding of clinics with name boards
  * Provision of family planning prescription booklets
  Interventions: Behavioral: FP Training and Technical Support
- Control Arm (No Intervention): the providers in the control group will continue to provide their services as usual with no exposure to intervention activities. After the end of the intervention period, providers that fall into control areas will be provided the same training.

INTERVENTIONS:
Behavioral: FP Training and Technical Support — Same as in Intervention arm description
  Arms: Intervention Arm

SUMMARY:
This study aims to generate evidence on the feasibility and effectiveness of engaging for-profit private sector family physicians and pharmacies to include family planning (FP) as a routine service in rural areas of Pakistan. The study will enlist family physicians and pharmacies in rural areas of Islamabad, Pakistan. Physicians will be randomly assigned to intervention and control groups. Those in intervention arm will received training on family planning and technical support for six months during the duration of the study, to evaluate the impact of training and support in expanding family planning coverage and impact.

DETAILED DESCRIPTION:
Pakistan has an overall national goal under the National Plan of Action on Population Growth and the national commitment for the international FP2030 goals to expand family planning services by raising Contraceptive Prevalence Rate (CPR) to 60 percent by 2030 in Pakistan . Based on the Population Council's earlier Landscape study of Family planning services, the total market approach has not been fully adopted in Pakistan (The Population Council, 2016). It called for the inclusion of the private sector and pharmacies to expand access to family planning services and commodities. Another study by the Council also explored the potential of including the private sector and proposed the case for engaging family physicians in family planning . The National Plan of Action on Population Growth's recommendation no. 2 calls for engaging the for-profit private sector, especially family physicians in efforts to expand family planning services . However, a review of evidence in 2020 noted that no determined effort was found to engage private physicians to provide family planning in a sustainable and for-profit model. Internationally, the involvement of the private sector in family planning has been proposed as a High Impact Practice (HIP). The ultimate goal of this study is to provide a model for a successful engagement of male family physicians and pharmacies in family planning and, thereby, expanding family planning services in rural areas to achieve universal access to FP. The engagement of for-profit (male) family physicians in the provision of FP services in linkage with pharmacies will combine three high-impact practices (HIPs) in family planning: (i) private sector engagement (ii) male participation in family planning (Khan, K & Sathar, Z, 2020) and (iii) integrating pharmacies in the health system.

This study aims to generate evidence on the feasibility and effectiveness of engaging for-profit private sector family physicians and pharmacies to include family planning (FP) as a routine service. It aims to fill the knowledge gap about the effectiveness of engaging private sector family physicians, and also the optimal approach of integrating family physicians' and pharmacies in Pakistan. Given that the lack of family planning services is particularly dire in rural areas, we situate the study in the rural areas of Islamabad. The study outcomes would provide evidence for advocacy for a sustainable model that can be scaled up to both rural and urban areas.

The study involves an intervention to test the feasibility of engaging male family physicians and pharmacies in expanding the provision of family planning services in the rural areas, on the basis of a review of previous studies, and discussions with a number of private providers, pharmacists, government officials and researchers, The impact of the intervention is to be tested through a randomized control study. The study will enlist family physicians and pharmacies in rural Islamabad Capital Territory (ICT) , who will give their written and informed consent to participate in the study. Physicians will be randomly assigned to intervention and control groups with equal chances of falling into each group.

* The intervention will provide male family physicians with training and technical support and integrates them with the nearest pharmacies or drug shops for vertical referrals. Technical support will include:
* Supportive supervision
* Peer-to-peer support
* Strengthening referrals for long-acting reversible contraceptives (LARC) and permanent methods
* Provision of information, education, and communication (IEC) material and LCD for display of visual material.
* Branding of clinics with signboards
* Provision of family planning prescription booklets The providers in the intervention group will receive the intervention package, the providers in the control group will continue to provide their services as usual with no exposure to intervention activities. After the end of the intervention period, providers that fall into control areas will be provided the same training. We hypothesize that the proposed intervention will enable male family physicians to provide information, counselling, family planning prescriptions, and referrals, as requested by clients and will result in increased uptake of contraceptive methods.

To evaluate intervention outcomes, baseline assessments in both intervention and control arms will obtain quantitative data from family physicians and pharmacies. We will assess our primary and secondary outcomes using the Management Information System (MIS) tool for obtaining routine service statistics data from clinics and contraceptive sales data from pharmacies. After 6 months of completing the intervention, end-line assessments will be conducted with family physicians in both intervention and control arms to measure changes in providers' KAP towards FP due to intervention. We will also interview family physicians in the intervention arm to get their feedback on the intervention's effectiveness and feasibility through in-depth interviews.

In addition, data on contraceptive availability and sales trends, monitoring stock positions, will be obtained from pharmacies, those nearest to; and linked with participating clinics, at the start, at 3 months, and at 6 months of intervention. The regular availability of contraceptives at the participating pharmacies will be ensured, and mechanisms to address declining stocks or stock outs would be addressed by linking with manufacturers and distributors and with health or population welfare department facilities if needed.

ELIGIBILITY:
Inclusion Criteria:

* Private clinics with a male family physician
* Male family physician working on a regular basis (3 or more days a week)
* Clinics located in Islamabad rural areas.

Exclusion Criteria:

* Clinics or facilities with specialized care (skin care, laser clinics, surgical clinics, among others)
* Clinics located in ICT urban areas
* Male family physicians working in a private clinic where a female medical doctor attends to patients during the same working hours.

Ages: 22 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study intends to engage male family physicians in family planning service provision in Pakistan. The gender identity is based on self-representation.
Enrollment: 76 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of family physicians successfully providing family planning services to their clients | 6-months
  the proportion of family physicians in the intervention arm compared to the control arm providing FP services to at least 10 per cent of their total clients during the intervention period.

SECONDARY OUTCOMES:
change in contraceptive uptake | 6-months
  2. Percentage point difference in contraceptive sales in pharmacies linked to clinics in the intervention arm as compared to the control arm.
change in number of FP clients | 6-months
  Estimate the average (mean) number of clients receiving FP services in the intervention group compared to the control group by the end of intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Ayaz Ahmed Baloch, Principal Investigator — Population Council
Locations (1):
- Population Council, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Federal and Provincial Task Force s, 2019, Action Plan (2019-24) for Implementation of Recommendations Approved by CCI Regarding Alarming Population Growth in Pakistan.
- [Background] The Population Council. 2016. Landscape Analysis of Family Planning Situation in Pakistan: Brief Summary of Findings. Islamabad: The Population Council
- [Background] Rehman Ashfaq and Malkani Anam. 2020. Best Bets for Accelerating Family Planning in Pakistan: The Case for Engaging Family Physicians and the for-Profit Private Sector. Islamabad: Population Research Center and the Population Council.
- [Background] Khan, K., & Sathar, Z. (2020). Best Bets for Accelerating Family Planning in Pakistan: Inducting men, sharing responsibility
- [Background] The Population Council. 2019. Improving Access to Family Planning Services through the Private Sector in Pakistan: A Stakeholder Analysis. Islamabad: The Population Council.
- [Background] Bradley, S.E & Shiras, T. Pharmacies and Drug Shops. Expanding contraceptive Choice and access in the private sector. Family Planning High Impact Practices2021